CLINICAL TRIAL: NCT03427151
Title: An Open-label Study of the Safety and Tolerability of Repeated Administration of a 200-mcg Dose of IPP-201101 Plus Standard of Care in Patients With Systemic Lupus Erythematosus
Brief Title: Study of Repeated Administration of a 200-mcg Dose of IPP-201101 Plus Standard of Care in Patients With Systemic Lupus Erythematosus
Acronym: IP-006
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ImmuPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPP-201101/006
Record Dates: First submitted 2017-12-08; First posted 2018-02-09 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — spliceosomal peptide P140

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IPP-201101 (Experimental): every 4 weeks
  Interventions: Drug: IPP-201101

INTERVENTIONS:
Drug: IPP-201101 — 200 mcg of IPP-201101 will be administered subcutaneously every 4 weeks for 24 weeks.

SUMMARY:
this study extension objective is to evaluate the safety and tolerability of a 200-mcg dose every 4 weeks for 24 weeks of IPP-201101 in patients with active systemic lupus erythematosus (SLE) who had participated in the main study IP-005.

ELIGIBILITY:
Inclusion Criteria:

* Patient had participated previously to study IP-005
* Written informed consent is obtained.
* Female and males receiving IPP-201101 and their female partners must use a highly effective contraceptive during treatment and for 30 days after discontinuation of study drug treatment.
* Women must be surgically sterile, 2 years postmenopausal, or, if of childbearing potential, use a highly effective method of contraception, Men and their partner must have highly effective accepted method of contraception. Single barrier/Double barrier and spermicides are not acceptable methods of contraception. Highly effective methods of contraception include, true abstinence, intrauterine device (IUD), or hormonal contraception associated with inhibition of ovulation (oral, transdermal, implanted, and injected), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner. True abstinence is defined when this is in line with the preferred and usual lifestyle of the subject." [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception]
* If the patient is using oral corticosteroids, the weekly cumulative dose must not exceed 80 mg of prednisone equivalent; the weekly dose must be stable over the 4 weeks preceding the 1st dose of study drug.
* If the patient is using antimalarials, methotrexate, leflunomide, mycophenolate mofetil (MMF), or azathioprine, the start date must be at least 3 months prior to the 1st dose of study drug, and the daily dose must be stable over the 4 weeks preceding the 1st dose of study drug.
* If the patient is not currently using corticosteroids, antimalarials, methotrexate, MMF, or azathioprine, the last dose (in case of previous use) must be at least 4 weeks prior to the 1st dose of study drug. For leflunomide, the stop date must be at least 8 weeks before the 1st dose of study drug unless an adequate cholestryamine washout has been performed. If cholestyramine washout is performed, the last use of leflunomide must be at least 4 weeks before the 1st dose of study drug.
* The patient must be willing and able to comply with study restrictions, to remain at the study center for the required duration during each study visit, and to return to the study center for the final assessment as specified in this protocol.

Criteria for Exclusion: Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* The patient has been treated with intramuscular or intravenous (iv) pulse steroids (ie, 250 to 1000 mg iv total daily dose of methylprednisolone) within 4 weeks of the 1st dose of study drug. The use of intra-articular steroids may be allowed after consultation with the medical expert.
* The patient has received tacrolimus, cyclosporin A, or iv immunoglobulins (IVIG) within 3 months of the 1st dose of study drug.
* The patient has received cyclophosphamide within 6 months prior to the 1st dose of study drug.
* The patient has been treated for SLE with agents such as fusion proteins, therapeutic proteins, or monoclonal antibodies or antibody fragments, within 6 months of the 1st dose of study drug.
* The patient has received B-cell depleting agents such as rituximab or belimumab or epratuzumab within one year of the 1st dose and has not yet normalized the B-cell count (ie, CD20+ B-cell count is less than normal range and the absolute lymphocyte count [ALC] is less than normal range).
* The patient has New York Heart Association (NYHA) Class III or IV congestive heart failure.
* The patient has an estimated glomerular filtration rate (eGFR) of less than 30 mL/min/1.73 m2 (via Modification of Diet in Renal Disease [MDRD] equation).
* The patient has an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value greater than 2 times the upper limit of the normal range (ULN) or a total bilirubin level greater than 1.5 times ULN.
* The patient has a planned immunization with a live or live attenuated vaccine within 3 months prior to administration of the 1st dose of study drug and for 3 months after administration of the last dose of study drug.
* The patient has any clinically significant abnormalities on ECG that are not related to SLE, as determined by the investigator. Patients with stable ECG changes without evidence of active cardiovascular disease may participate at the discretion of the investigator and medical monitor.
* The patient has an ongoing active systemic infection requiring treatment or a history of severe infection, such as hepatitis or pneumonia, in the 3 months prior to administration of the 1st dose of study drug. Less severe infections in the 3 months prior to administration of the 1st dose of study drug are permitted at the discretion of the investigator and medical monitor.
* The patient has any concomitant medical condition unrelated to SLE that may interfere with his or her safety or with evaluation of the study drug, as determined by the investigator.
* The patient has a history of a medical condition other than SLE that has required treatment with oral corticosteroids in excess of 80 mg of prednisone equivalent/week within 3 months of the 1st dose of study drug.
* The patient has a positive test result for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab).
* The patient has a known positive history of antibodies to human immunodeficiency virus (HIV) or HIV disease or other immunosuppressive state (eg, agammaglobulinemia, etc).
* The patient has a history of alcohol or substance dependence or abuse (with the exception of nicotine),according to the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, Fourth Edition, Text Revision (DSM-IV-TR), within 3 months of the screening visit or has current substance abuse.
* The patient has a history of severe allergic reactions to or hypersensitivity to any component of the study drug.
* The patient has undergone or is undergoing treatment with another investigational drug for the treatment of lupus within 6 months prior to the 1st dose of study drug or has received any other investigational drug for any other condition within 4 weeks prior to the 1st dose of study drug except for IPP-201101
* The patient is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* The patient is unlikely to comply with the study protocol or is unsuitable for any other reason, as judged by the investigator or medical monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events throughout the study | 7 months
  all adverse events will be coded using MedDRA and the sverity will be graded according to the modified WHO toxicity Criteria and they will be determined by the Investigator to be treatment related. The incidence of adverse events will be summarized using descriptive statistics by system organ classe and preferred term.
Clinical laboratory test results at each visit during the treatment extension period | 7 months
  Summary statistics for laboratory tests will be presented at baseline and at each visit.The severity of select laboratory resuts will be graded accroding the Modified WHO Toxicity Criteria.
Body weight measurements at each visit during the treatment period | 7 months
  The incidence of clinically significant abonormal values will be summarized using descriptive statistics.
Temperature measurements at each visit during the treatment period | 7 months
  The incidence of clinically significant abonormal values will be summarized using descriptive statistics.
Pulse measurements at each visit during the treatment period | 7 months
  The incidence of clinically significant abonormal values will be summarized using descriptive statistics.
Systolic and diastolic blood pressures measurements at each visit during the treatment period | 7 months
  The incidence of clinically significant abonormal values will be summarized using descriptive statistics.
2-lead electrocardiogram (ECG) findings at week 28 (or final assessment) | 7 months
  Any ECG finding that is judged by the investigator as a clinically significant change (worsening) compared to a baseline value will be considered an adverse event coded using MedDRA
Physical examination findings, at specified time points at each visit during the treatment extension period | 7 months
  Body system (General appearance, Skin, HEENT (Head, eyes, ears, nose, throat), Lymph Nodes, Thyroïd, Musculo-skeletal / Extremities, Cardiovascular, Lungs, Abdomen, Neurological) findings that is judged by the investigator as a clinically significant change (worsening) compared to a baseline value will be considered an adverse event coded using MedDRA
Concomitant medication usage throughout the study extension | 7 months
  All concomittant medication will be coded using the WHO Drug dictionnary. The incidence of concomittant medications will be sumamrized using descriptive statistics by therapeutic class and preferred terms category.

SECONDARY OUTCOMES:
the effect in the Clinical SLEDAI-2K total score by at final visit compared to initial visit | at week 28
  The SLEDAI 2K is a validated objective measure that assesses disease activity within the last 28 days before completion of the index. It is a global index and includes 24 weighted clinical and laboratory variables. The SLEDAI-2K clinical score is the calculated score without inclusion of the points that may be contributed by having a psoitive titer fr anti-dsdna Ab or decreased serum complement level. The SLEDAI-2K clinical score (sum of 22 scores) ranges from 0 to 101.
remission of the disease (i.e reduction of clinical SLEDAI-2K score to 0) | at week 28

CONTACTS AND LOCATIONS:
Locations (14):
- United States (4):
  - WALLACE, Los Angeles, California
  - East Bay Rheumatology Medical, San Leandro, California
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Innovative Health Research, Las Vegas, Nevada
- Czechia (2):
  - Revmatologie s.r.o., Brno
  - Revmatologický ústav v Praze, Prague
- France (2):
  - GHR Mulhouse Sud-Alsace, Mulhouse
  - CHU de la Réunion, Saint-Denis
- Germany (2):
  - Schlosspark-Klinik Berlin, Berlin
  - Clinic for Rheumatology and Internal Medicine, Freiburg im Breisgau
- Hungary (2):
  - University of Debrecen Medical Center Department of Clinical Immunology, Debrecen
  - Mentaház Magánorvosi Központ Kft., Székesfehérvár
- CAP Research, Phoenix, Mauritius
- Latin Clinical Trial Center, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No